CLINICAL TRIAL: NCT05139056
Title: A Phase I Study of Multiple Doses of Neural Stem Cell-Based Oncolytic Virotherapy (NSC-CRAd-S-pk7) Administered Intracerebrally to Patients With Recurrent High-Grade Gliomas
Brief Title: Multiple Intracerebral Doses of Neural Stem Cell-Based Virotherapy (NSC-CRAd-S-pk7) for the Treatment of Recurrent High-Grade Gliomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22338; NCI-2022-10170 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22338 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-11-22; First posted 2021-12-01 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Currently Only Enrolling Glioblastoma Patients at First Recurrence
Keywords: Recurrent glioblastoma, oncolytic virus, neural stem cells, first recurrence
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (NSC-CRAd-S-pk7) (Experimental): Patients undergo standard surgical resection, and during surgery the first dose of study agent is injected into the wall of the resection cavity. Patients then receive three additional doses every week or every two weeks (depending on when they enroll in the study) via a catheter that was placed during surgery
  Interventions: Biological: Neural Stem Cells-expressing CRAd-S-pk7; Procedure: Resection

INTERVENTIONS:
Biological: Neural Stem Cells-expressing CRAd-S-pk7 — Given intracerebrally
  Other Names: CRAd-S-pk7 loaded NSCs; NSC-CRAd-S-pk7; NSC-CRAd-S-pk7 Virotherapeutic; NSCs loaded with CRAd-S-pk7; SC-CRAd-Survivin-pk7
Procedure: Resection — Undergo surgical resection
  Other Names: Intracerebral administration of NSC-CRAd-S-pk7 via intracavitary catheter; Removal of CSF samples via a catheter placed in the lateral cerebral ventricle

SUMMARY:
This phase I trial studies the safety of giving multiple intracerebral doses of NSC-CRAd-S-pk7 to treat patients with glioblastoma at first recurrence. NSC-CRAd-S-pk7 consists of neural stem cells that can target glioblastoma cells and carry a virus, which can kill cancer cells. Giving multiple doses of NSC-CRAd-S-pk7 may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the recommended maximum tolerated number of cycles (MTC) of intracavitary (ICT) administered neural stem cell-expressing CRAd-S-pk7 (NSCCRAd-S-pk7) for phase II testing based on dose-limiting toxicities (DLTs), the overall toxicity profile, and activity in patients with recurrent high-grade glioma (HGG).

II. Describe and compare the weekly dosing schedule (Treatment Schedule 4) to an every 2 week dosing schedule (Treatment Schedule 4a) of intracerebrally administered NSC-CRAd-S-pk7 based on DLTs, the overall toxicity profile, and activity in patients with glioblastoma at first recurrence.

III. Determine the recommended phase 2 dose schedule based on the overall toxicity profile, and activity in patients with recurrent high grade gliomas

SECONDARY OBJECTIVES:

I. I. Assess for evidence of biologic activity (cytotoxicity and anti-tumor immune responses) in posttreatment tissue samples.

II. Assess for the presence of NSC and/or CRAd-S-pk7 in post-treatment tissue samples.

III. Assess for possible development of antibody and T cell responses to the NSCs and/or CRAd-S-pk7 in CSF and blood.

IV. Assess for evidence of possible migration of NSCs and/or CRAd-S-pk7 outside of the brain and if so, determine if viral shedding is occurring.

V. Determine the persistence and intracerebral distribution of the NSCs and/or CRAd-S-pk7 whenever permission is given to perform a brain autopsy on a study participant.

VI. Estimate the rates of disease response, progression-free survival at 6 months (PFS6mo) and overall survival at 9 months (OS9mo) for all study participants and separately for the cohorts of glioblastoma patients at first recurrence treated at the MTC administered once a week or every 2 weeks.

VII. Identify a molecular signature of vulnerability for predicting which glioma patients will benefit most from treatment with NSC-CRAd-S-pk7.

VIII. Describe and compare changes in immunosuppressive and immunostimulatory cytokines in CSF from study participants enrolled to Treatment Schedules 4 and 4a.

IX. Assess for the presence of exhausted T cell phenotypes in CSF samples and compare the degree of T cell exhaustion in study participants enrolled to Treatment Schedules 4 and 4a.

OUTLINE:

Patients undergo standard surgical resection, and during surgery the first dose of study agent is injected into the wall of the resection cavity. Patients then receive three additional doses every week or every two weeks via a catheter placed during surgery. A second catheter is placed in the cerebral ventricle to obtain serial samples of CSF for correlative studies. Two weeks after the last dose of study agent is administered, study participants undergo a second surgical procedure to remove the catheters and obtain post-treatment tissue samples for analysis.

FINANCIAL ASSISTANCE:

There is funding to help with the cost of transportation, lodging, and meals for participants who qualify for financial assistance.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be age >= 18 years
* Patient has a Karnofsky performance status of >= 70%
* Patient has a life expectancy of >= 3 months

  * When determining the maximum tolerated number of treatment cycles (MTC): patient has a histologically confirmed diagnosis of a grade 3 or 4 glioma (eg., glioblastoma, grade 4 astrocytoma, grade 3 astrocytoma, grade 3 oligodendroglioma). (This part of the study has been completed).
  * When enrolling to Treatment Schedules 4 and 4a: patient has glioblastoma at first recurrence.
* Imaging studies show evidence of recurrent, supratentorial tumor(s).
* Patient's high-grade glioma has recurred or progressed after prior treatment with brain radiation and temozolomide
* The patient must be in need of surgery for tumor resection
* Based on the neurosurgeon's judgment, there is no anticipated physical connection between the post-resection tumor cavity and the cerebral ventricles
* Absolute neutrophil count (ANC) of >= 1000 cells/mm^3
* Platelet count >= 100,000 cells/mm^3
* Total bilirubin =< 2.0 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 4 times the institutional upper limit of normal
* Serum creatinine =< the institutional upper limit of normal
* At least 2 weeks from taking the last dose of a targeted agent
* At least 4 weeks from the last dose of bevacizumab For temozolomide, an interval of 23 days is required from the last dose administered if the patient was recently treated with adjuvant temozolomide, consisting of temozolomide daily for 5 days, repeated every 28 days.
* At least 2 weeks from taking the last dose of a targeted agent.
* At least 4 weeks from the last dose of bevacizumab.
* All significant toxicities from previous anticancer therapy must have stabilized to a new baseline or resolved.
* All participants must have the ability to understand and the willingness to sign a written informed consent.
* The effects of this treatment on a developing fetus are unknown. Therefore, female patients of childbearing potential and sexually-active male patients or who are able to impregnate their partner, must agree to use an effective method of contraception while participating in this study. Patients of childbearing potential must have a negative pregnancy test =< 2 week prior to registration.

Exclusion Criteria:

* Patient has multi-focal disease.
* Patient is receiving radiation, chemotherapy, or another investigational agent.
* Patient has had prior therapy with neural stem cells.
* Patient has not recovered from any toxicity (> grade 1) of prior therapies, except alopecia.
* Patient is unable to undergo a brain MRI.
* Patient has chronic or active viral infections of the central nervous system (CNS).
* Patient has a coagulopathy or bleeding disorder.
* Patient has an uncontrolled illness including ongoing or active infection.
* Patient has another active malignancy.
* Patient is pregnant or breastfeeding.
* A patient has a serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the safety monitoring requirements and completion of treatment according to this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-08-07 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days post removal of Rickhams
  Assessed using the Common Terminology Criteria for Adverse Events version 5.0.
Progression-free survival (PFS) | From the time of surgery to the event date of progression, assessed at 6 months]
  Will estimate the rate 90% confidence interval (CI) for PFS at 6 months and use Kaplan Meier methods to estimate median PFS for all study participants as well as for the cohorts of glioblastoma (GBM) participants at first recurrence who will be treated with 4 doses of NSC-CRAd-S-pk7 given once a week or every two weeks.

SECONDARY OUTCOMES:
Neural Stem Cells-expressing CRAd-S-pk7 (NSC-CRAd-S-pk7) immunogenicity | Up to 30 days post removal of Rickhams
NSC-CRAd-S-pk7 migration within the brain | Up to 30 days post removal of Rickhams
  Neural stem-cells and/or free viral particles will be assessed in samples of post-treatment tissue samples.
NSC-CRAd-S-pk7 migration outside the brain | Up to 30 days post removal of Rickhams
  4. Neural stem-cells and/or free viral particles will be assessed in samples of CSF, peripheral blood, urine, oral and rectal mucosa (via swabbing), and skin at the injection site (also via swabbing).
Disease response | Up to 2 years
  Response Assessment in Neuro-Oncology Criteria will be used to assess response on brain magnetic resonance imaging in all study participants who receive at least 80% of the planned doses of study treatment. Disease response will be similarly assessed for the cohorts of GBM participants at first recurrence who will be treated with 4 doses of NSC-CRAD-S-pk7 once a week or every two weeks.
Overall survival (OS) | From time of surgery to date of death, assessed at 9 months
  Will estimate the rate 90% CI for OS at 9 months and use Kaplan Meier methods to estimate median OS for all study participants as well as for the cohorts of GBM participants at first recurrence who will be treated with 4 doses of NSC-CRAd-S-pk7 once a week or every two weeks.
Changes in HSPG and survivin expression | Baseline up to 2 years
  Changes in survivin expression by immunohistochemistry IHC in pre- and post-treatment tissue to see if there is a relationship with disease response.
Changes in immune cell populations | Baseline up to 2 years
  Changes in immune cell populations in the tumor microenvironment in pre- and post-treatment tumor tissue samples will be assessed by Vectra Spectral Imaging.
Changes in tumor growth | Baseline up to 2 years
  Develop a biomathematical model for predicting tumor response to study treatment.
Assessed using multiplex immunoassays in cerebrospinal fluid (CSF) samples and RNA-sequencing in CSF, peripheral blood, and tumor tissue samples. | Up to 30 days post removal of Rickhams

CONTACTS AND LOCATIONS:
Overall Officials: Jana L Portnow, MD, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - Standford University, Stanford, California
  - Northwestern University, Chicago, Illinois
  - Wake Forest University, Winston-Salem, North Carolina